CLINICAL TRIAL: NCT07184281
Title: Effectiveness of School-Based Time-Restricted Eating for the Prevention and Control of Obesity in Children: A Cluster-Randomized Controlled Trial
Brief Title: Effectiveness of School-Based Time-Restricted Eating for the Prevention and Control of Obesity in Children
Acronym: SCHOOL-TRE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Soochow University (Other)
Collaborators: Soochow University (Other)
Responsible Party: Principal Investigator, Xiaoyan Shi, Clinical Professor, Children's Hospital of Soochow University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SCHOOL-TRE; SYW2025048 (Other Grant/Funding Number: Suzhou Municipal Science and Technology Bureau)
Record Dates: First submitted 2025-08-18; First posted 2025-09-19 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Childhood Obesity; Childhood Obesity Pevention
Keywords: childhood obesity; school-based intervention; time-restricted eating; cluster randomized trial
MeSH Terms: conditions — Pediatric Obesity; Intermittent Fasting

STUDY DESIGN:
Intervention Model Description: cluster randomized trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TRE group (Experimental): Based on the current health education model, the subjects in the experimental group were administered for 12 hours of TRE.
  Interventions: Behavioral: 12-hour time-restricted eating; Behavioral: health education
- Control group (Active Comparator): The current health education model is adopted, that is, health education is carried out in accordance with the "Guiding Outline for Health Education in Primary and Secondary Schools".
  Interventions: Behavioral: health education

INTERVENTIONS:
Behavioral: 12-hour time-restricted eating — Based on the current health education model, the subjects in the experimental group were administered for 12 hours of TRE. Carry out the propaganda and education of the 12-hour TRE feeding mode, the core content is that the eating time window is limited to 12 hours/day, the last meal is no later than 19:00, the study subjects can freely choose the eating time window, do not restrict energy intake during eating, and during the fasting period, they are allowed to drink non-calorie, sugar-free drinks (water, tea, coffee). Record the time of eating every day.
  Arms: TRE group
Behavioral: health education — The current health education model is adopted, that is, health education is carried out in accordance with the "Guiding Outline for Health Education in Primary and Secondary Schools".

SUMMARY:
Childhood obesity has become a major global public health challenge. Obesity can not only affects children's physical and mental health during childhood but may also persist into adulthood, significantly increasing the risk of cardiovascular disease. Therefore, effective prevention and control of childhood obesity can shift the prevention window forward and promote the prevention of cardiovascular disease. Recently, time-restricted eating (TRE) has gained attention in adult studies for its feasibility, as it involves "time control without calorie restriction," demonstrating weight loss effects comparable to energy restriction and higher feasibility. Here, the investigators designed a school-based cluster randomized controlled trial to investigate the effectiveness of 12-hour TRE in preventing and controlling childhood obesity. Schools were randomly assigned to either the intervention group or the control group, and participants were recruited from each school at the class level, ensuring that each group included at least 690 children. The control group received routine health education, while the intervention group received 12-hour TRE in addition to routine health education. After a 9-month intervention period (one academic year), the two groups will be compared in terms of weight management and childhood obesity prevalence.

DETAILED DESCRIPTION:
Childhood obesity has become a major global public health challenge. With rapid economic development, the prevalence of childhood obesity in China has risen from 0.1% in 1985 to 7.3% in 2024. Childhood obesity not only affects children's physical and mental health during childhood but may also persist into adulthood, significantly increasing the risk of cardiovascular disease. Therefore, effective prevention and control of childhood obesity can shift the prevention window forward and promote the prevention of cardiovascular disease. The age distribution of childhood obesity shows that the peak incidence occurs between 7 and 12 years of age, making this a critical period for prevention and control. During this stage, children are in school, spending half their time there, and exhibit strong behavioral plasticity. Interventions based on school settings may be an effective approach to preventing and controlling childhood obesity. Previous experimental studies have shown that comprehensive school-based interventions (primarily including reducing overeating, high-energy diets, and sedentary behavior, while increasing physical activity) can significantly reduce BMI and childhood obesity prevalence, but their feasibility is limited. Recently, time-restricted eating (TRE) has gained attention in adult studies for its feasibility, as it involves "time control without calorie restriction," demonstrating weight loss effects comparable to energy restriction and higher feasibility. Therefore, the investigators hypothesize that a 12-hour TRE program implemented in schools may enhance the prevention and control of childhood obesity, but there is currently a lack of empirical evidence, particularly regarding its preventive effects on childhood obesity. Here, the investigators designed a school-based cluster randomized controlled trial to investigate the effectiveness of 12-hour TRE in preventing and controlling childhood obesity. Schools were randomly assigned to either the intervention group or the control group, and participants were recruited from each school at the class level, ensuring that each group included at least 690 children. The control group received routine health education, while the intervention group received 12-hour TRE in addition to routine health education. After a 9-month intervention period (one academic year), the two groups will be compared in terms of weight management and childhood obesity prevalence.

ELIGIBILITY:
Eligibility criteria for schools:

1. The principal agrees to accept the randomization process and adhere to the study protocol;
2. The total number of fourth-year students in the school must be more than 50;
3. Schools that have not implemented or plan to implement obesity prevention interventions;
4. Non-boarding schools, Ethnic minority schools, or specialty schools;
5. Schools that have no clear plans to relocate or close within the next 2 years;

Eligibility criteria for classes:

1. Class teachers are willing and actively involved in home-school liaison;
2. Class sizes should be between 30 and 60 students;
3. The class consists of fourth-grade students;
4. Classes that have no clear plan to merge or cancel in the next 2 years;

Exclusion criteria for students:

All students in the selected classes will be the subject of the study after signing the informed consent, unless they have the following circumstances:

1. Individuals with a history of heart disease, high blood pressure, diabetes, tuberculosis, asthma, hepatitis or nephritis;
2. Individuals with secondary obesity: obesity due to endocrine disorders or side effects of medications;
3. Individuals with abnormal growth and development, such as dwarfism, gigantism, etc;
4. Individuals with physical deformities, including severe scoliosis, chicken breasts, claudication, significant O-leg/X-shaped legs;
5. Individuals with limited athletic ability who are unable to participate in school physical activities;
6. Individuals who have lost weight by inducing vomiting or taking medication in the past 3 months;
7. Individuals who have undergone prior bariatric surgery;
8. Individuals with mental disorders or intellectual developmental disabilities, as well as aphasia;
9. Individuals who have taken medications that affect appetite or weight within three months (e.g., antipsychotics, hypnotics, weight loss medications, insulin);
10. Individuals who have plans to transfer within 2 years;

Ages: 8 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1380 (Estimated)
Dates: Start 2025-09-26 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
change in BMI-Z score | From enrollment to the end of treatment at 9 months
  change in BMI-Z score from baseline

SECONDARY OUTCOMES:
change in the prevalence of overweight or obesity | From enrollment to the end of treatment at 9 months.
  change in the prevalence of children with a BMI-Z score over 2 from baseline
chang in BMI | From enrollment to the end of treatment at 9 months.
  change in BMI from baseline
change in waist-to-hip ratio | From enrollment to the end of treatment at 9 months.
  change in waist-to-hip ratio from baseline
change in blood pressure | From enrollment to the end of treatment at 9 months.
  change in blood pressure from baseline
change in eating behavior | From enrollment to the end of treatment at 9 months.
  Change in eating behavior from baseline. The Child Eating Behavior Questionnaire (CEBQ), designed to assess children's eating scale styles, will be used in our study. It is a parent-report measure comprised of 35 items, each rated on a five-point Likert scale that ranges from never to always. It is made up of eight scales: Food responsiveness, Emotional over-eating, Enjoyment of food, Desire to drink, Satiety responsiveness, Slowness in eating, Emotional under-eating, and Food fussiness. The instrument is ideal for use in research investigating the early precursors of eating disorders or obesity.
change in physical activity | From enrollment to the end of treatment at 9 months.
  Change in physical activity from baseline. The Physical Activity Questionnaire for Adolescents (PAQ-A), a self-report scale designed for use with school students, will be used to assess the physical activity in our study. It contains eight items intended to capture adolescents' recollections of their physical activity over the preceding 7 days. The first and last of the PAQ-A's eight items each contain a number of subitems from which a mean is initially calculated, and those two means are added to responses on the other six items to obtain a total from which the mean is calculated to produce a composite score ranging from 1 to 5, with higher scores indicating greater physical activity. A ninth question seeks information about anything that would have prevented respondents from engaging in their "normal physical activities" during the previous week.
change in life quality | From enrollment to the end of treatment at 9 months.
  Change in life quality from baseline. The Quality of Life Scale for Children and Adolescents (QLSCA) is a Chinese version of the quality of life Scale for Children and Adolescents, consisting of 49 items for measuring 13 dimensions of students' lives, such as their relationships with teachers and parents, partnership with fellow students, learning abilities and attitudes, self-perception, physical well-being, negative emotions, attitudes towards homework, living environment convenience, social activities, sports capacity, self-satisfaction, and other unspecified factors. The QLSCA uses a five-point Likert-type scale to measure either frequency or intensity, with a recall period of two weeks. Scores were calculated for each dimension, with higher scores indicating a better quality of life.

OTHER OUTCOMES:
longterm effect | From enrollment to 1 year after intervention.
  change in BMI-Z score at 1 year after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoyan Shi, PhD, Principal Investigator — Children's Hospital of Soochow University
Locations (2):
- China (2):
  - Children's Hospital of Soochow University, Suzhou, Jiangsu
  - Wujiang Center for Disease Prevention and Control, Suzhou, Jiangsu

IPD SHARING:
Plan to Share IPD: No
The unidentified patient data can be shared.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-08-10): https://cdn.clinicaltrials.gov/large-docs/81/NCT07184281/Prot_SAP_000.pdf